CLINICAL TRIAL: NCT01088035
Title: A Phase II Multi-Institutional Trial of Focal Radiotherapy With Concomitant Carboplatin as a Radiosensitizer and the Prospective Analysis of Survivin, an Inhibitor of Apoptosis, as a Biomarker in Children With Newly Diagnosed Non-Metastatic Ependymoma and Minimal Residual Disease Post-Operatively
Brief Title: Carboplatin as a Radiosensitizer in Treating Childhood Ependymoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Jason Fangusaro, Attending, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMH 09C4
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Ependymoma
Keywords: Childhood ependymoma; Ependymoma; Survivin
MeSH Terms: conditions — Ependymoma; Familial ependymoma | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carboplatin (Experimental)
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Carboplatin — Patients will receive daily carboplatin as a radiation sensitizer prior to radiation each day.

SUMMARY:
This is a phase II study evaluating the feasibility of concurrent carboplatin given with focal radiation therapy in children age 12 months to < 21 years with newly diagnosed localized ependymoma who have no or minimal residual disease post-operatively (< 0.5 cm). The hypothesis is that utilizing carboplatin as a radiosensitizer is feasible and tolerable and may improve event-free survival (EFS) and minimize local recurrences as compared to historic controls. Following a neurosurgical resection and staging, patients who meet the eligibility criteria will receive standard fractionated radiation therapy at doses of 54 to 59.4 Gy to the primary site depending upon age. All patients will receive 35 mg/m²/day of carboplatin prior to each fraction of radiotherapy. Although significant neutropenia is not anticipated, G-CSF will be administered per study guidelines during radiation if neutropenia occurs. All patients will be followed for toxicity, response (resolution of residual disease) and event-free survival (EFS). Patients' tumor sample, blood and cerebro-spinal fluid (CSF) will also be prospectively evaluated to quantify the level of Survivin, a known inhibitor of apoptosis, via immunohistochemistry, Western Blot Analysis (in tumor tissue) and ELISA (in blood and CSF). The feasibility of obtaining these levels prospectively and in real time will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be enrolled before treatment begins.
* Patients must be ≥ 12 months and < 22 years of age at the time of diagnosis.
* The target tumors are primary brain non-metastatic (M0) ependymomas tumors. Patients must have histologic verification of an ependymoma at diagnosis. Patients with the following world health organization (WHO) diagnoses will be eligible for this study:Ependymoma (Subtypes: cellular, papillary, clear cell and tanycytic) and Anaplastic Ependymoma
* Life expectancy of ≥ 8 weeks.
* Newly diagnosed ependymoma and must not have had any prior chemotherapy or radiotherapy.
* All patients must have:

  * A pre-operative MRI scan of the brain with and without contrast. NOTE: CT scans are NOT sufficient for study eligibility since radiation therapy planning and responses will be based on MRI scans only.
  * Post-operative head MRI scan with and without contrast (preferably within 72 hours post-operatively).
  * Spinal MRI (T-1 weighted imaging with and without gadolinium) is required within 28 days of surgery if done post-operatively and within 14 days of surgery if done pre-operatively. For posterior fossa tumors, pre-operative MRI scans are preferred because surgically induced inflammation/blood can be difficult to distinguish from tumor.
  * Lumbar CSF cytology examination obtained between 7 and 31 days following surgery.
  * Adequate bone marrow function, defined as:
  * Peripheral absolute neutrophil count (ANC) >1500/μL
  * Platelet count ≥ 100,000/μL (transfusion independent)
  * Hemoglobin ≥ 10.0 gm/dl (may receive RBC transfusions)
  * Adequate renal function defined as:
  * Serum creatinine < 1.5 times the upper limit of normal based on the patient's age, or creatinine clearance greater than 60 ml/min/1.73 m² corrected for age and body surface area.
  * Adequate liver function defined as:
  * Total bilirubin <1.5 x the institutional normal
  * SGOT (AST) or SGPT (ALT) <2.5 x institutional normals.
* Patients must begin chemoradiotherapy within 56 days of definitive surgery.
* All patients and/or their parents or legal guardians must sign a written informed consent
* Patients must provide assent as per local IRB guidelines (if applicable).
* Patients and/or their families must consent to the mandatory biology studies, including serum Survivin levels, CSF Survivin levels, paraffin-embedded tissue and fresh-frozen tissue when available.
* Karnofsky/Lansky scoring greater than 50.
* Corticosteroid supportive care is permissible at the clinician's discretion prior to and during chemo-radiotherapy.
* Anti-seizure medication support is permitted as necessary and at the treating physician's discretion.

Exclusion:

* Prior chemotherapy or prior radiotherapy
* Patients who are pregnant or breast feeding, or patients (male or female) not employing adequate contraception. Acceptable means of birth control include IUD, oral contraceptive, subdermal implant, a condom with a contraceptive sponge or suppository or abstinence.
* Patients who are unable to undergo MR imaging
* Patients with evidence of metastatic disease on spine MRI or CSF sampling
* Patients with post-operative residual tumor > 0.5 cm, unless a repeat surgery is performed making the residual tumor less than 1.5 cm². Note: Timing for enrollment and initiation of therapy will begin after second surgery if a repeat surgery is performed.

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2010-04; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Measure the EFS of newly diagnosed non-metastatic ependymoma patients treated with a combination of daily carboplatin as a radiosensitizer and conformal radiotherapy. | 3 years
Explore the tolerability, feasibility and toxicities associated with daily carboplatin as a radiosensitizer in patients with newly diagnosed non-metastatic ependymoma receiving focal fractionated radiotherapy. | 1 year
  Tolerability and toxicity will be measured by documenting the toxicities associated with this treatment using the current CTCAE version 4.0. The feasibility of this therapy will be measured by observing the ability to finish therapy without delays and the ability to receive daily carboplatin and radiation in the time alloted by the study (within 4 hours) on a daily basis. Delays in therapy will be documented in an effort to define both tolerability and feasibility.

SECONDARY OUTCOMES:
Explore the overall survival (OS) in patients with newly diagnosed non-metastatic ependymoma treated with this regimen. | 3 years
Evaluate the feasibility of quantifying Survivin expression in primary ependymoma tumor, blood and CSF samples in a prospective fashion. | 6 months
Explore trends or relationships between Survivin expression (in tumor, blood and CSF samples) and tumor histology. | 3 years
Explore trends or relationships between Survivin expression (in tumor, blood and CSF samples) and patient responses. | 3 years
Explore trends or relationships between Survivin expression (in tumor, blood and CSF samples) and survival outcomes. | 3 years
Explore trends or relationships between Survivin expression (in tumor, blood and CSF samples) tumor recurrences. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Fangusaro, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Rachel Altura, MD, Principal Investigator — Brown University
Locations (1):
- Children's Memorial Hospital, Chicago, Illinois, United States